CLINICAL TRIAL: NCT06140550
Title: Prospective, Multicenter, Randomized Controlled Clinical Trial to Evaluate the Effectiveness and Safety of Biolimus-coated Intracranial Balloon Dilation Catheter Treatment of Patients With Symptomatic Intracranial Atherosclerotic Stenosis
Brief Title: Clinical Trial of Biolimus-coated Intracranial Balloon Dilation Catheter
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bochang (Industry)
Collaborators: Xuanwu Hospital, Beijing (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); First People's Hospital of Hangzhou (Other); Jinan Central Hospital (Other); The Affiliated Hospital of Qingdao University (Other); Beijing Geriatric Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TP-NS-036
Record Dates: First submitted 2023-11-14; First posted 2023-11-20 (Actual); Last update posted 2023-11-20 (Actual); Status verified 2023-11

CONDITIONS: Intracranial Atherosclerotic Stenosis
Keywords: Intracranial balloon; stenosis
MeSH Terms: conditions — Constriction, Pathologic

STUDY DESIGN:
Intervention Model Description: Ratio of control group to test group 1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Device: Drug balloon dilated
- Control group (Experimental)
  Interventions: Device: balloon dilated

INTERVENTIONS:
Device: Drug balloon dilated — Through the expansion after the balloon is in place,Release drugs on the surface of the balloon and improve the blood perfusion of nerve vessels to treat stenosis
  Arms: Experimental group
Device: balloon dilated — Through the expansion after the balloon is in place, improve the blood perfusion of nerve vessels to treat stenosis.
  Arms: Control group

SUMMARY:
This test took the target lesion restenosis rate 6 months after the operation as the main endpoint to verify the effectiveness of the intracranial balloon expansion catheter of Biolimus coating. After completing the follow-up 6 months after the operation, a clinical summary report was issued for the registration application of the product, and on this basis, 12 months of postoperative follow-up was carried out to evaluate the mid-term curative effect.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old;
* Symptomatic intracranial artery stenosis, and the degree of visual stenosis of target blood vessels under intracranial angiography is 70~99%(WASID method);

Exclusion Criteria:

* Target blood vessels are seriously calcified and distorted, and it is difficult to put the interventional instruments in place or recover;
* Ischemic cerebral infarction occurred 3 weeks before surgery;
* Cerebral hemorrhage 3 months before operation;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
6-month target lesion restenosis rate | 6-month